CLINICAL TRIAL: NCT06695208
Title: Histomorphometric and Radiographic Assessment of Bone After Socket Preservation Using Biodentin Versus Xeno Graft for Socket Preservation of Single Rooted Mandibular Teeth: Randomized Clinical Trial
Brief Title: Socket Preservation Using Biodentin Versus Xeno Graft for Single Rooted Teeth
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maxim Salib Todry Gerges, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD_CU_2024-01-26
Record Dates: First submitted 2024-11-08; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Socket Perservation
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- biodentine group (Experimental)
  Interventions: Drug: Biodentine
- xeno graft group (Active Comparator)
  Interventions: Drug: Biodentine

INTERVENTIONS:
Drug: Biodentine — biodentine used in socket preservation

SUMMARY:
socket preservation using biodentin versus xeno graft for single rooted mandibular teeth

DETAILED DESCRIPTION:
after extraction of single rooted mandibular teeth the socket will be filled with xeno graft or biodentine and the socket will be closed using gel foam and sutures then CBCT will be taken to measure bone width after 6 months of healing CBCT will be taken again to measure the difference in bone width and a core biopsy will be taken followed by implant placement

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex with badly decayed tooth indicated for extraction
* The ages of the patients ranged from 25 to 50 years.
* Patients with healthy systemic condition (Medically free)
* Adequate inter-arch space for placement of the implant prosthetic part.
* Good oral hygiene
* Cooperative patients who are willing to commit for 6 months follow up

Exclusion Criteria:

* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Poor oral hygiene and motivation.
* Smokers
* Patient with medical condition that contraindicates surgical procedures
* Pregnant or nursing.
* Substance abuse.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or parafunctional habits severe bruxism or clenching.
* Active infection or severe inflammation in the area intended for implant placement.
* Patients on medication that may interfere with healing (corticosteroids, bisphosphonate, Chemo/radio therapy).

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
radiographic assessment to calculate bone width in millimeters after socket preservation in mandibular single rooted teeth using cone beam computed tomography | 6 months postoperative
  calculation of bone width gain in millimeters in extraction socket in mandibular single rooted teeth using cone beam computed tomography.

SECONDARY OUTCOMES:
Histomorphometric analysis of bone after socket preservation in mandibular single rooted teeth harvested by trephine bur | 6 months postoperative
  assessment of bone quality from extraction socket that were preserved bone will be harvested using trephine bur followed by implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Starch-Jensen T, Vitenson J, Deluiz D, Ostergaard KB, Tinoco EMB. Lateral Alveolar Ridge Augmentation with Autogenous Tooth Block Graft Compared with Autogenous Bone Block Graft: a Systematic Review. J Oral Maxillofac Res. 2022 Mar 31;13(1):e1. doi: 10.5037/jomr.2022.13101. eCollection 2022 Jan-Mar. PMID 35574210
- [Result] Gerritsen AE, Allen PF, Witter DJ, Bronkhorst EM, Creugers NH. Tooth loss and oral health-related quality of life: a systematic review and meta-analysis. Health Qual Life Outcomes. 2010 Nov 5;8:126. doi: 10.1186/1477-7525-8-126. PMID 21050499
- [Result] Henry PJ. Tooth loss and implant replacement. Aust Dent J. 2000 Sep;45(3):150-72. doi: 10.1111/j.1834-7819.2000.tb00552.x. PMID 11062933
- [Result] Iorio-Siciliano V, Blasi A, Nicolo M, Iorio-Siciliano A, Riccitiello F, Ramaglia L. Clinical Outcomes of Socket Preservation Using Bovine-Derived Xenograft Collagen and Collagen Membrane Post-Tooth Extraction: A 6-Month Randomized Controlled Clinical Trial. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):e290-e296. doi: 10.11607/prd.2474. PMID 28817143
- [Result] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Result] Rajasekharan S, Martens LC, Cauwels RGEC, Anthonappa RP. Biodentine material characteristics and clinical applications: a 3 year literature review and update. Eur Arch Paediatr Dent. 2018 Feb;19(1):1-22. doi: 10.1007/s40368-018-0328-x. Epub 2018 Jan 25. PMID 29372451
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- See also: Lateral Alveolar Ridge Augmentation with Autogenous Tooth Block Graft Compared with Autogenous Bone Block Graft: a Systematic Review — https://pubmed.ncbi.nlm.nih.gov/35574210/
- See also: Tooth loss and oral health-related quality of life: a systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/21050499/
- See also: Tooth loss and implant replacement — https://pubmed.ncbi.nlm.nih.gov/11062933/
- See also: Clinical Outcomes of Socket Preservation Using Bovine-Derived Xenograft Collagen and Collagen Membrane Post-Tooth Extraction: A 6-Month Randomized Controlled Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/28817143/
- See also: Preservation of alveolar bone in extraction sockets using bioabsorbable membranes — https://pubmed.ncbi.nlm.nih.gov/9776033/
- See also: Biodentine™ material characteristics and clinical applications: a 3 year literature review and update — https://pubmed.ncbi.nlm.nih.gov/29372451/
- See also: Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study — https://pubmed.ncbi.nlm.nih.gov/12956475/